CLINICAL TRIAL: NCT04848753
Title: A Phase III Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate Perioperative Toripalimab (JS001) Combined With Neoadjuvant Chemotherapy in Patients With Resectable Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma
Brief Title: Perioperative Toripalimab (JS001) Combined With Neoadjuvant Chemotherapy in Patients With Resectable Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS001-042-III-ESCC
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Resectable Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma
MeSH Terms: interventions — Cisplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Active Comparator): Toripalimab combined with cisplatin and paclitaxel
  Interventions: Combination Product: Toripalimab combined with cisplatin and paclitaxel
- Control Group (Placebo Comparator): Placebo combined with cisplatin and paclitaxel
  Interventions: Combination Product: Placebo combined with cisplatin and paclitaxel

INTERVENTIONS:
Combination Product: Toripalimab combined with cisplatin and paclitaxel — Specified doses on specified days.
  Arms: Experimental Group
Combination Product: Placebo combined with cisplatin and paclitaxel — Specified doses on specified days.
  Arms: Control Group

SUMMARY:
This is a randomized, placebo-controlled, multi-center, double-blinded, Phase III study to determine the efficacy and safety of patients with locally advanced squamous cell carcinoma of the thoracic esophagus treated with perioperative immunotherapy combined with neoadjuvant chemotherapy versus placebo combined with neoadjuvant chemotherapy.

ELIGIBILITY:
Patients must fulfill all of the following inclusion criteria to be eligible for enrollment in this study:

1. Histologically confirmed locally advanced (T1N1-3M0 or T2-3N0-3M0) squamous cell carcinoma of the thoracic esophagus (per the 8th Edition of UICC-TNM Classification);
2. No suspicious cervical lymph node metastasis on cervical contrast-enhanced CT; no systemic metastasis from radiological examination;
3. Expected to be achievable to conduct R0 resection.

Patients must not enter this study if any of the following exclusion criteria is fulfilled:

1. Having malignant tumors other than esophageal carcinoma within 5 years prior to randomization;
2. Combined with other inoperable condition;
3. Previous serious allergy to chemotherapeutic agents (paclitaxel or cisplatin) or any monoclonal antibody;
4. Combined with other conditions unsuitable for participation in this study as judged by investigators.

Other protocol defined Inclusion/exclusion criteria could apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 663 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2027-05-12 (Estimated); Study Completion 2027-05-12 (Estimated)

PRIMARY OUTCOMES:
To compare IRC-assessed events-free survival (EFS) in 2 arms | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed approximately up to 60 months

SECONDARY OUTCOMES:
pathologically complete remission (pCR) rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed approximately up to 60 months
  To compare the percentage of patients who achieved pCR in the 2 arms, pCR rate was defined as the percentage of subjects who achieved a complete pathological response (PCR)
Investigator-assessed EFS according to RECIST v1.1 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed approximately up to 60 months
  To compare Investigator-assessed events-free survival (EFS) in patients with locally advanced squamous cell carcinoma of the thoracic esophagus treated with perioperative immunotherapy combined with neoadjuvant chemotherapy versus placebo combined with neoadjuvant chemotherapy.
Overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed approximately up to 60 months
  To compare Overall survival in patients with locally advanced squamous cell carcinoma of the thoracic esophagus treated with perioperative immunotherapy combined with neoadjuvant chemotherapy versus placebo combined with neoadjuvant chemotherapy.
1-year OS rate | from randomization to death from any cause at 1 year
  To compare 1-year OS rates in patients with locally advanced squamous cell carcinoma of the thoracic esophagus treated with perioperative immunotherapy combined with neoadjuvant chemotherapy versus placebo combined with neoadjuvant chemotherapy
3- year OS rate | from randomization to death from any cause at 3 year
  To compare 3-year OS rates in patients with locally advanced squamous cell carcinoma of the thoracic esophagus treated with perioperative immunotherapy combined with neoadjuvant chemotherapy versus placebo combined with neoadjuvant chemotherapy
5- year OS rate | from randomization to death from any cause at 5 year
  To compare 5-year OS rates in patients with locally advanced squamous cell carcinoma of the thoracic esophagus treated with perioperative immunotherapy combined with neoadjuvant chemotherapy versus placebo combined with neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute; Yongtao Han, Principal Investigator — Sichuan Cancer Hospital and Research Institute; Yan Zheng, Principal Investigator — Henan Cancer Hospital; Keneng Chen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (48):
- China (48):
  - The Firest Affiliated Hospital of bengbu Medical College, Bengbu, Anhui
  - Anhui provincial hospital, Hefei, Anhui
  - The Second Hospital of anhui Medical University, Hefei, Anhui
  - Jiangmen central Hospital, Jiangmen, Guangdong
  - Shenzhen people's hosptial, Shenzhen, Guangdong
  - The fourth hospital of hebei medical university, Shijiazhuang, Hebei
  - Anyang Cancer Hospital, Anyang, Henan
  - The First Affiliated Hospital of xinxiang Medical University, Xinxiang, Henan
  - Henan provincial pepples hospital, Zhengzhou, Henan
  - The first affilated hospital of zhengzhou university, Zhengzhou, Henan
  - Hunan provincial cancer hospital, Changsha, Hunan
  - China-Japan Union hosptial of Jilin university, Changchun, Jilin
  - The first affiliated hospital of jinzhou medical university, Jinzhou, Niaoning
  - Shanxi provincial cancer hosptial, Taiyuan, Shanxi
  - Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Hwa Mei Hospital,University of Chinese Academy of sciences, Ningbo, Zhejiang
  - Taizhou hospital of zhejiang province, Taizhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The General Hospital of People's Liberation Army, Beijing
  - Heping Hospital Affiliated to changzhi Medical College, Changzhi
  - Sichuan Cancer Hospital & Institute, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - 3201 Hospital, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hanzhou
  - harbin medical university Cancer Hospital, Harbin
  - Anhui Provincial Cancer Hospital, Hefei
  - Huai'an First People's Hospital, Huai'an
  - The Affiliated Hospital of jining Medical University, Jining
  - The First Affiliated Hospital of nanchang University, Nanchang
  - Jiangsu Cancer Hospital, Nanjing
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Zhongshan Hospital Fudan University, Shanghai
  - Shantou University Cancer Hospital, Shantou
  - Liaoning cancer hospital& Institute, Shenyang
  - Shengjing Hospital of China Medical University, Shenyang
  - The first Hospital of china Medical University, Shenyang
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Hubei Cancer Hospital, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Zhongshan Hospital Affiliated to Xiamen University, Xiamen
  - Xinyang central Hospital, Xinyang
  - The Affiliated Hospital of xuzhou Medical University, Xuzhou
  - Yantai yuhuangding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou